CLINICAL TRIAL: NCT00223548
Title: MESNA Zur Prophylaxe Der Kontrastmittel-Induzierten Nephropathie
Brief Title: MESNA for Prevention of Acute Deterioration of Renal Function Following Contrast Agent Application
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Ulm (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: A119/2002
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2002-09

CONDITIONS: Chronic Renal Insufficiency; Serum Creatinine Concentration; Contrast Media Exposition
Keywords: prophylaxis; contrast-induced nephropathy; mesna; acute renal failure
MeSH Terms: conditions — Renal Insufficiency, Chronic; Acute Kidney Injury | interventions — Mesna

INTERVENTIONS:
Drug: sodium 2-mercaptoethane sulfonate

SUMMARY:
The purpose of this study is to determine wether Mesna could prevent contrast-induced nephropathy

DETAILED DESCRIPTION:
Contrast-induced nephropathy remains a common complication of radiographic precedures. Pretreatment with Mesna (Sodium 2-mercaptoethane sulfonate) in combination with sodium chloride is more protective than sodium chloride alone in animal models of acute renal failure.

The aim of this study is therefore to determine laboratory and clinical benefit of MESNA, as an adjunct to saline hydration, in patients with known renal impairment receiving contrast media.

ELIGIBILITY:
Inclusion Criteria:

* stable chronic renal insufficiency
* serum creatinine concentration > 1,5 mg/dl

Exclusion Criteria:

* Dialyzed patients
* patients with acute renal failure
* received iodinated contrast media within 7 days before study entry
* known allery to Mesna, pregnancy, and administration of dopamine, mannitol or N-acetylcysteine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106
Dates: Start 2002-10; Study Completion 2004-12

PRIMARY OUTCOMES:
Contrast-agent associated nephrotoxicity was defined as an increase in serum creatinine concentration >0.5 mg/dl (44 umol/l) of the baseline value 48 h after administration of the contrast media.

SECONDARY OUTCOMES:
Need for dialysis after the administration of contrast media.

CONTACTS AND LOCATIONS:
Overall Officials: Frieder Keller, M.D., Principal Investigator — Division of Nephrology, University Hospital Ulm; Frieder Keller, M.D., Principal Investigator — Division of Nephrology, University Hospital of Ulm
Locations (1):
- Division of Nephrology, University of Ulm, Ulm, Germany